CLINICAL TRIAL: NCT06939933
Title: Effect of Aquatic Exercises on Muscle Strength and Quality of Life in Children With Sickle Cell Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Eman Samir Shaltout, eman samir shaltout, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-462
Record Dates: First submitted 2025-04-09; First posted 2025-04-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Anemia in Children
Keywords: aquatic exercises; sickle cell anemia; rehabilitation; quality of life; muscle power; children
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Intervention study model Parallel assignment The study will include 50 spastic children suffering from sickle cell anemia ( age 6 to 10 years and divided into 2 randomized subgroups.
  Group (A): Will receive aquatic exercised in addition to the designed physical
  Physical program :
  Group (B): Will receive the designed physical therapy program only.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (A) (Experimental): aquatic exercised in addition to the designed physical
  Interventions: Other: aquatic exercise in addition to physical exercise
- group (B) (Experimental): designed physical therapy program only
  Interventions: Genetic: designed physical exercises only

INTERVENTIONS:
Other: aquatic exercise in addition to physical exercise — Aquatic exercise refers to the use of water that facilitates the application of established therapeutic interventions, including stretching, strengthening, joint mobilization, balance and gait training and endurance training. Water has been throughout history for a variety of purposes including ; physical therapy, rehabilitation and sport. There activities are made possible by water's special qualities and the influence of these attributes on humans.
  Hydrotherapy is one of the most popular forms of complementary therapies that help in the treatment of children with disabilities. It is known to provide an opportunity to the children to do easier exercise. It also improves .
  Physical therapy and tailored exercise programs can help improve muscle strength, endurance, and overall physical function in children with SCA. Such programs need to be carefully designed to avoid triggering pain crises while promoting physical health and improving quality of life.
  Arms: group (A)
Genetic: designed physical exercises only — Physical therapy and tailored exercise programs can help improve muscle strength, endurance, and overall physical function in children with SCA. Such programs need to be carefully designed to avoid triggering pain crises while promoting physical health and improving quality of life (Ballas et al., 2010).
  benefit from anaerobic activity patterns (Dougherty et al., 2018). A study to examine maximal muscle strength and peak power in children with sickle cell anemia found that maximal muscle strength and peak power are significantly less in children with sickle cell anemia compared to the control group
  Arms: group (B)

SUMMARY:
Sickle cell anemia is a global public health disorder that aﬀects millions of people across the globe. It is an inherited autosomal recessive hemoglobin condition caused by a beta-globin gene mutation that results in an aberrant sickle cell hemoglobin molecule with glutamic acid replaced by valine at position six of the beta-globin chain.

Sickle cell anemia is a hereditary illness characterized by persistent microvascular blockage by sickle-shaped cells, chronic hemolytic anemia, and tissue destruction. Red-cell dehydration, hypoxemia, metabolic acidosis, and hyperthermia are typical vaso-occlusive triggers.

Children with sickle cell anemia frequently have poor growth and nutritional status, increased protein turnover, decreased lean body mass, and elevated resting and lower activity energy expenditures.

These clinical findings present a problem for recommending exercise when taken as a whole, while engaging in physical activity increases the chance of issues like a "painful episode,". Children with sickle cell anemia miss out on the favorable health effects of regular physical activity, such as the growth of lean body mass, strength, and fitness.

Vaso-occlusive events are recurring and prevalent in sickle cell anemia-related morbidity. Patients also have a higher chance of developing central nervous system conditions such cerebral vasculopathy and overt and covert stroke. It has been noted that the pathophysiological symptoms of SCA decrease skeletal muscle function. In fact, it has been demonstrated that individuals with SCA have diminished forearm and respiratory muscular maximal strength as well as peak locomotory muscle power.

Vaso-occlusion, chronic hemolytic anemia, and vasculopathy form the core of sickle cell anemia pathophysiology and result in both acute and chronic consequences that have a significant negative influence on quality of life QoL. Even though clinical care for children with SCA has significantly improved in developed countries over the past few decades, children and adolescents with SCA still have a lower quality of life than their peers due to painful vaso-occlusive crises, frequent hospital admissions, and lengthy hospital stays.

Generic and disease-specific measures of quality of life have been developed and validated in chronic illnesses to evaluate the influence of health on functional domains such physical and mental well-being, exhaustion, pain, social engagement, relationships, and emotional distress. Examples include the Child Health Questionnaire, Pediatric Quality of Life Sickle Cell Disease Module PedsQL SCD, and Patient-Reported Outcomes Measurement Information System PROMIS, all of which have been used to study SCA and have revealed various degrees of quality-of-life impairment, primarily in the United States.

Health-related quality of life refers to the patient's assessment of how his or her well-being and level of functioning, in comparison to the perceived ideal, are influenced by personal health. A health-related quality of life assessment often considers physical, social, and emotional functioning in addition to academic and occupational performance.

Studies on the quality of life for people with SCA have significantly risen during the previous five years. Measurement of health-related quality of life is beneficial for many reasons. Health-related quality of life can be used to measure the efficacy and effectiveness of treatment interventions, to predict outcomes and resource use, and to direct therapy. More importantly, the measurement of health-related quality of life aids in understanding the burden of disease that patients experience.

DETAILED DESCRIPTION:
Aquatic exercise refers to the use of water that facilitates the application of established therapeutic interventions, including stretching, strengthening, joint mobilization, balance and gait training and endurance training. Water has been throughout history for a variety of purposes including ; physical therapy, rehabilitation and sport. There activities are made possible by water's special qualities and the influence of these attributes on humans.

Hydrotherapy is one of the most popular forms of complementary therapies that help in the treatment of children with disabilities. It is known to provide an opportunity to the children to do easier exercise. It also improves .

Provides then with the ability to do movements with fun especially among children who enjoy doing training activities when moving on the ground is difficult for them.

Aquatic exercises are especially helpful in cases where a land -based exercises , program is not possible due to the intensity of pain, decreased bone density, disability or other factors. All of these conditions can make it uncomfortable or painful to exercises on a hard or even padded surface or while standing. Water provides a much gentler welcoming environment.

This review of literature provides a clear understanding of the current concepts under the following subheadings:

1- Sickle cell anemia

1. Definition
2. Incidence
3. Pathophysiology
4. Clinical features
5. Complications
6. Management 2- Muscle strength and sickle cell anemia 3- Health related quality and sickle cell anemia

   1. Sickle cell anemia

      1. Definition It is an inherited hemoglobinopathy caused by a single amino acid substitution at the sixth residue of the beta (β)-globin subunit, which results in the production of the characteristic Hemoglobin S. It is induced by β-globin gene mutation and influences millions of people worldwide.

         The disease primarily affects the development of red blood cells, resulting in the formation of hemoglobin -S (is an abnormal type of hemoglobin which causes RBCs to become sickle-shaped and inflexible, this is usually the most severe form of the disease. These abnormal cells clump together in the arteries blocking blood flow to various organs and hence cause various complications. Sickle cell anemia is considered a genetic disorder, distinguished by Vaso-occlusive crises (VOCs) and hemolytic anemia.
      2. Incidence This disease is most common in India, sub-Saharan Africa, and the Mediterranean area, but is also detected in wider Americas and Europe. About 100,000 people in the United States and millions more across the world suffer from sickle cell anemia, SCD occurs among about 1 out of every 365 Black or African American births. SDC occurs among about 1 out of every 16,300 Hispanic American births. About 1 in 13 Black or African American babies is born with sickle cell trait. The incidence of sickle cell disease increased from 4.62 to 4.65% globally, reaching 5.46 million individuals in 2021.

         Sadly, the illness kills about 300,000 children under the age of five every year-five times more than other causes of death. To put things in perspective, there were roughly 4,400 sickle cell-related fatalities worldwide in 2021. Nevertheless, the Global Burden of Disease Study 2023 (GBD 2023) appears to have significantly underestimated these figures, as it was unable to fully capture their scope.

         In the Caribbean and sub-Saharan Africa, the impact is even more profound due to the high prevalence of the trait in these regions. For instance, the Caribbean saw an increase in sickle cell disease-related mortality from 425,000 to 515,000.

         These figures underscore the critical need for enhanced data collection and reporting methods to ensure accurate tracking and management of sickle cell disease globally.
      3. Pathophysiology Hemoglobin S displays biochemical characteristics): when hemoglobin S is deoxygenated, it crystallizes together with related polymers, causing the structure of red blood cells to distort (the recognizable sickle shape). Increased red blood cell density, Hemoglobin S polymerization that causes red blood cells to become irreversibly sickled, a fall in cell ion and water content (cell dehydration), and cyclic deoxygenation are all related to cyclic deoxygenation.

         First, ischemic/reperfusion damage is brought on by microvascular blockages in capillaries and small vessels due to the sickle cells' enhanced adhesiveness. Vaso-occlusive events in microcirculation are the result of a complicated scenario that is still only partially understood. This scenario involves interactions between various cell types, including leukocytes, platelets, plasma factors, abnormally activated endothelial cells, dense red blood cells, and reticulocytes. the local reduction in nitric oxide bioavailability. Extra- and intra-vascular hemolytic disease are caused by either the red blood cells' increased stiffness and resulting in reduced deformability, which results in either their evacuation by macrophages (liver or spleen) or their destruction inside the circulation.

         When thymine replaces adenine in the beta globin gene's sixth codon, valine (a hydrophobic amino acid) is produced instead of glutamic acid, which is hydrophilic, leading in SCA. Despite that, all people with sickle cell anemia have the same genetic mutation; each patient's clinical history is very different.
      4. Clinical features The symptoms of SCA can vary from person to another and can change over time. The early symptoms are yellowish skin color (jaundice), whites of eyes (icterus), extreme tiredness, painful swelling of hands and feet (dactylitis).

         There are recent studies that mention that there are three most frequent symptoms including fatigue, bone aches, and headaches. 67% rated the severity of symptoms with fatigue, in the array of "severe" to "worst imaginable Likert score 5-7. In case of bone aches and headache, the severity was valued by 67% and 54% of patients. Psychological symptoms were also predominant, with 38% and 39% of patients suffering anxiety and depression.
      5. Complications Some complications may be systemwide (affect many parts of the body at the same time), others affect specific parts.

         According to Pinto et al., 2019, Complications affecting the whole body may include:
         * Acute pain crisis: Also called Vaso-occlusive crisis It occurs without warning, when sickled cells lock blood flow. People describe that pain as sharp, intense, stabbing, or throbbing. Common areas affected by that pain include the abdomen, chest, lower back, arms, or legs.
         * Vitamin deficiency: People with SCA are at a high risk for nutrient and vitamin deficiency specially vitamin D, omega 3, vitamin C, and zinc that can also causes a crisis or complications.
         * Chronic long-term pain: Chronic pain is common, but it can be hard to describe. It is always different from crisis pain the results from organ damage.
         * Delayed growth and puberty: Because of the resulting anemia, children with SCA may grow and develop more slowly than their peers.
         * Infections: Because of the damaged spleen, the risk for certain infections is higher in patients with sickle cell anemia. Including chlamydia, H. influenza type B, salmonella, and staphylococcus.
         * Joint problems sickling in the hip bones and, less commonly, the shoulder joint, knees, and ankles can reduce oxygen flow and result in a condition called avascular or aseptic necrosis which severely damage the joints. The symptoms include pain, problems with walking and joint movement.
         * Blood clots: Change in how the blood travels through blood vessels can result in blood clots. Swelling of arms or legs, pain or tenderness not caused by injury, sudden shortness of breath, weakness in specific areas of the body, changes in thinking maybe some signs of blood clotting.
         * High blood pressure: People with sickle cell anemia can develop high blood pressure, increase the workload of the heart and blood vessels, and worsen high-risk complications like stroke and kidney diseases.
         * Serious anemia complications: Severe anemia in a newborn or a child who has a sickle cell anemia may be a result of one of two conditions; Aplastic crisis: is usually caused by Parvovirus B19 infection which is also called slapped chick syndrome. Parvovirus B19 can cause the bone marrow to stop producing new red blood cells for a while leading to severe anemia. Or splenic sequestration crisis: most commonly occurs in newborns and children who have sickle cell anemia.

         Patients with SCA who are exposed to malaria are at a higher risk of sickle cell crisis and death Williams and Obaro, 2011 and have a greater danger of pneumococcal disease especially children younger than 5 years, diarrheal disease, and infections in bone associated with Vaso-occlusive crisis.

         The Comprehensive Sickle Cell Centers Clinical Trial Consortium exhibits the occurrence of different complications such as sickle cell pain and asthma, as well as cumulative age noticeably lessened scores in the vitality domain (i.e., were allied with elevated incidence of fatigue.
      6. Management of sickle cell anemia Current management of SCA focuses primarily on the maintenance of health and treatment of acute and chronic complications. Several important modalities such as hydroxyurea therapy and blood transfusion have been found to boost patient outcomes.

      Hydroxyurea therapy reduces the frequency of vasooclusive crisis and acute splenic sequestration crisis, acute chest syndrome therapy reducing the need for blood transfusions and associated hospitalizations, while stem cell transplantation is the intervention that most likely to be curative in nature. However, this option is often associated with several complications.

      Hematopoietic stem-cell transplantation and gene therapy can cure SCA but require significant healthcare resources and can have severe health consequences. As of 2021, only six centers in Africa offer transplantation, while 215 centers in the USA can perform transplants National Marrow Donor Program.

      High-resource settings may provide better care, but there is room for improvement in quality care and further research is needed to understand the factors contributing to negative outcomes in SCA.
   2. Muscle strength and sickle cell anemia Child's overall health, play activity, and quick movement in an emergency, it is crucial to maintain optimal muscle function throughout childhood. To perform something, anaerobic exercise is frequently required. Furthermore, kids often perform brief bursts of vigorous movement while they are playing. Because of this, a child's daily life can benefit from anaerobic activity patterns.

A study to examine maximal muscle strength and peak power in children with sickle cell anemia found that maximal muscle strength and peak power are significantly less in children with sickle cell anemia compared to the control group. Children with SCA frequently have poor growth and nutritional status, increased protein turnover, decreased lean body mass, and elevated resting and lower activity energy expenditures. There is a severe lack of empirically supported information regarding anerobic performance among the few exercise research comparing children with sickle cell anemia to healthy children because most of these studies concentrated on aerobic performance.

Children with SCA often exhibit reduced muscle strength and endurance, which can further compromise their physical functioning and overall quality of life. Impact on Muscle Function: The chronic hemolytic anemia characteristic of SCA leads to reduced oxygen delivery to tissues, including muscles. This, combined with recurrent Vaso-occlusive crises, can contribute to muscle weakness and reduced exercise tolerance.

Objective measures of muscle strength, such as hand-held dynamometry, have shown that children with SCA have significantly lower muscle strength compared to healthy controls. These findings underscore the importance of incorporating muscle strength assessment and targeted interventions in the management of children with SCA.

Physical therapy and tailored exercise programs can help improve muscle strength, endurance, and overall physical function in children with SCA. Such programs need to be carefully designed to avoid triggering pain crises while promoting physical health and improving quality of life.

Sickle cell anemia significantly impacts the health-related quality of life and muscle strength in children. Addressing these challenges requires a multidisciplinary approach that includes medical management, physical rehabilitation, and psychological support to improve outcomes and enhance the quality of life for children living with this chronic condition. Future research should continue to explore innovative interventions and support mechanisms to mitigate the impact of SCA on children's physical and emotional well-being.

Assessment of muscle strength Muscle strength testing is a crucial part of diagnosing children with neurological and musculoskeletal dysfunctions. Objective muscle strength measurements provide baseline data and information about the pace of improvement. Commonly used clinical techniques for assessing muscle strength include manual muscle testing, Lafayette dynamometry, and hand-held dynamometry.

Manual muscle test Grades for a manual muscle test are recorded as numeric ordinal scores ranging from zero (0), which represents no discernable muscle activity, to five (5), which represents a maximal or best possible response or as great a response as can be evaluated by a manual muscle test. The numeric 0 to 5 system of grading is the most used for muscle strength scoring convention across health care professions. Each numeric grade can be paired with a word grade that describes the test performance in qualitative, but not quantitative, terms.

Lafayette handheld dynamometer Lafayette Hand-Held Dynamometer (L-HHD) is a valid and proven assessment tool used for objectively quantifying muscle strength. It is the ideal instrument for documenting medical necessity for tracking the progress during rehabilitation or a strength training program.

The Lafayette HHD features a wide range of customizable options for data storage, force overtime graphs, preset test times, and force thresholds. It includes three stirrups with an algometer attachment, users guide, battery charger, sanitary covers, and carrying case. Clinically, it was evaluated for children aged 4-17 years, it was concluded that it is valid and reliable in assessing muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* The children are assigned aged from 6-10 years.
* Both genders were included.
* They were able to follow instructions and understand commands.
* Children were free from orthopedic deformities in the upper and lower limbs.
* Children were not practicing any kind of sports.
* Children must have a normal body mass index (BMI) in relation to their ages.

Exclusion Criteria:

* Children with neurological, musculoskeletal, and cardiopulmonary diseases limit their movement.
* Children with cognitive disorders.
* Children suffering from auditory impairment that limit him or her from answering the questions.
* Children with vaso occlusive crises.
* Children who have another disease associated with SCA.
* Children who had recent blood transfusion.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
assessing hand grip strength | 3 months
  Hand-held dynamometer for assessing hand grip strength
assess weight | 3 months
  The Calibrated floor Health scale was used to assess weight
assessing Lower limb, trunk muscles strength. | 3 months
  3- Lafayette dynamometer for assessing Lower limb and trunk muscles strength.
determine the child's standing height in centimeters (cm). | 3 months
  The calibrated floor health scale was used to determine the child's standing height in centimeters (cm).
assessing Health related quality of life | 3 months
  4- Pediatric quality of life inventory 3.0 generic for assessing Health related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Eman samir shaltout, Tanta, Egypt